CLINICAL TRIAL: NCT03382405
Title: A Phase 1, Randomized, Observer-Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of Cytomegalovirus Vaccines mRNA-1647 and mRNA-1443 When Administered to Healthy Adults
Brief Title: Safety, Reactogenicity, and Immunogenicity of Cytomegalovirus Vaccines mRNA-1647 and mRNA-1443 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: mRNA-1647/mRNA-1443-P101
Record Dates: First submitted 2017-12-06; First posted 2017-12-22 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Cytomegalovirus Infection
Keywords: cytomegalovirus vaccine; mRNA-1647; mRNA-1443; Moderna
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — mRNA-1647 cytomegalovirus vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- mRNA-1647 (Experimental)
  Interventions: Biological: mRNA-1647
- mRNA-1443 (Experimental)
  Interventions: Biological: mRNA-1443
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: mRNA-1647 — Escalating dose levels
  Arms: mRNA-1647
Biological: mRNA-1443 — Escalating dose levels
  Arms: mRNA-1443
Other: Placebo — Saline
  Arms: Placebo

SUMMARY:
This clinical study will assess the safety, reactogenicity and immunogenicity of mRNA-1647 and mRNA-1443 cytomegalovirus vaccines in healthy adults

ELIGIBILITY:
Inclusion Criteria:

* Agrees to comply with the study procedures and provides written informed consent
* 18 to 49 years of age
* Body mass index between 18 and 35 kg/m2
* In good health based on medical history, physical examination, vital sign measurements and laboratory safety tests performed prior to initial study vaccination
* Negative urine pregnancy test at the Screening visit and the day of each vaccination for females of childbearing potential
* Female subjects must either be of non-childbearing potential or use acceptable methods of contraception from at least 30 days prior to enrollment and through 3 months following last vaccination
* Male subjects must agree to practice adequate contraception for 30 days prior to the first vaccination and through 3 months following the last vaccination
* Willing to comply with the requirements of the protocol (eg, complete Diary Cards, return for follow-up visits, be available for safety phone calls)

Exclusion Criteria:

* Any ongoing, symptomatic acute or chronic illness requiring medical or surgical care
* A history of malignancy in the last 10 years
* If female and of childbearing potential, is pregnant or lactating, has not adhered to an adequate contraception method from at least 30 days before study entry, or does not plan to do so for at least 3 months after the last vaccination.
* Abnormal screening safety laboratory test results including liver enzyme tests
* Administration of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the first dose of study vaccine or has plans for administration during the study period
* Prior administration of investigational agent using lipid nanoparticle formulations
* A positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus types 1 or 2 antibodies
* A positive test result for drugs of abuse
* Chronic administration of potentially hepatotoxic drugs or have other medical conditions that affect the liver (eg, alcohol abuse)
* A history of idiopathic urticaria
* Plans for administration or has been administered a vaccine within the period from 30 days before through 30 days after each study vaccination, with the exception of any licensed influenza vaccine administered ≥15 days before or after any study vaccination
* Any chronic administration of an immunosuppressant or other immune modifying drug
* Prior administration of immunoglobulins and/or any blood products within the 3 months before the first study vaccine or has plans for administration during the study period
* Any known or suspected immune-mediated disease or immunosuppressive condition as determined by medical history and/or physical examination
* A history of hypersensitivity or serious reactions to previous vaccinations
* Any bleeding disorder considered a contraindication to IM injection or blood draw
* Any acute illness or fever at screening
* Any condition that, in the opinion of the investigator, would pose a health risk to the subject if enrolled or could interfere with evaluation of the study drug or interpretation of study results
* Dose-escalation phase only, is seropositive for CMV at the Screening visit
* Donation of blood or blood products > 450 mL within 30 days of dosing.
* Is an immediate family member or household member of study personnel
* A history of seizure disorder for which anticonvulsants are currently prescribed

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 181 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2020-10-28 (Actual)

PRIMARY OUTCOMES:
Frequency of solicited AEs (local and systemic reactogenicity events) | 7 days following each dose administration
Frequency of unsolicited adverse events | 29 days following each dose administration
Frequency of medically-attended AEs, adverse events of special interest (AESI), and serious adverse events (SAE) | one year following the last dose administration
Frequency of clinical laboratory adverse events | 1 month following the last dose administration

SECONDARY OUTCOMES:
Titers of anti-CMV neutralizing antibodies against epithelial cell infection measured by neutralization assay in comparison with baseline sample | 6 months following the last dose administration
Titers of anti-CMV neutralizing antibodies against fibroblast cell infection measured by neutralization assay in comparison with baseline sample | 6 months following the last dose administration
Titers of vaccine antigen-specific IgG antibodies as measured by ELISA assay in comparison with baseline sample | 6 months following the last dose administration
Frequencies of vaccine antigen-specific CD4 and CD8 T cells secreting interferon gamma as determined by ELISPOT | 6 months following the last dose administration

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Research Centers of America, Hollywood, Florida
  - Advanced Clinical Research, Meridian, Idaho
  - Optimal Research, Peoria, Illinois
  - Johnson County Clinical Trials, Lenexa, Kansas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu K, Hou YJ, Makrinos D, Liu R, Zhu A, Koch M, Yu W-H, Paila YD, Chandramouli S, Panther L, Henry C, DiPiazza A, Carfi A. Characterization of humoral and cellular immunologic responses to an mRNA-based human cytomegalovirus vaccine from a phase 1 trial of healthy adults. J Virol. 2024 Apr 16;98(4):e0160323. doi: 10.1128/jvi.01603-23. Epub 2024 Mar 25. PMID 38526054
- [Derived] Fierro C, Brune D, Shaw M, Schwartz H, Knightly C, Lin J, Carfi A, Natenshon A, Kalidindi S, Reuter C, Miller J, Panther L. Safety and Immunogenicity of a Messenger RNA-Based Cytomegalovirus Vaccine in Healthy Adults: Results From a Phase 1 Randomized Clinical Trial. J Infect Dis. 2024 Sep 23;230(3):e668-e678. doi: 10.1093/infdis/jiae114. PMID 38478705
- [Derived] Hu X, Karthigeyan KP, Herbek S, Valencia SM, Jenks JA, Webster H, Miller IG, Connors M, Pollara J, Andy C, Gerber LM, Walter EB, Edwards KM, Bernstein DI, Hou J, Koch M, Panther L, Carfi A, Wu K, Permar SR. Human Cytomegalovirus mRNA-1647 Vaccine Candidate Elicits Potent and Broad Neutralization and Higher Antibody-Dependent Cellular Cytotoxicity Responses Than the gB/MF59 Vaccine. J Infect Dis. 2024 Aug 16;230(2):455-466. doi: 10.1093/infdis/jiad593. PMID 38324766